CLINICAL TRIAL: NCT04014920
Title: Non-invasive Ventilation Following Extubation (Prophylactic) to Prevent Extubation Failure in Critically Obese Patients: a Prospective, Randomized, Multicenter Study
Brief Title: Non-invasive Ventilation Following Extubation (Prophylactic) to Prevent Extubation Failure in Critically Obese Patients
Acronym: EXTUB-OBESE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19_0068
Record Dates: First submitted 2019-07-09; First posted 2019-07-10 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Ventilation; Intensive Care Unit
MeSH Terms: conditions — Obesity; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxygen Group (Active Comparator): Patient will receive standard oxygenotherapy
  Interventions: Device: Oxygen group
- NIV Group (Experimental): Patient will receive non invasive ventilation
  Interventions: Device: NIV Group

INTERVENTIONS:
Device: Oxygen group — The control group will receive oxygen (first randomization), HFNO oxygen or standard oxygen (second randomization)
  Arms: Oxygen Group
Device: NIV Group — The experimental group will receive NIV (first randomization) alternated with HFNO or standard oxygen (second randomization)
  Arms: NIV Group

SUMMARY:
Mechanical ventilation is the first artificial support used in intensive care. After a period of invasive mechanical ventilation, patients should be separated from the ventilator (weaning period of mechanical ventilation). If weaning and extubation (removal of the tracheal tube) are successful in approximately 80 to 90% of resuscitation patients, 10 to 20% will develop acute respiratory failure (ARF) in the days following extubation. Obesity concerns 20 to 30% of resuscitation admissions in France. The pathophysiological changes in the obese patient explain the over-risk of desaturation and ARF in the post-extubation period. In order to decrease the incidence of extubation failure (need for reintubation within 48-72h post-extubation) of the most fragile patients, it is recommended in intensive care unit to prophylactically use various ventilatory support strategies and / or oxygenation, among which noninvasive ventilation (NIV) and oxygen therapy, which can be administered in two ways: High-Flow Humidified Nasal Oxygen Therapy (HFNO) or standard oxygen therapy. These strategies have never been compared in the obese post-extubation critically ill patient. Our hypothesis is that NIV is superior to oxygen to prevent the development of ARF in obese extubated patients in intensive care unit.

DETAILED DESCRIPTION:
Mechanical ventilation is the first artificial support used in intensive care unit (ICU). After a period of invasive mechanical ventilation, patients should be separated from the ventilator (weaning period of mechanical ventilation). If weaning and extubation (removal of the tracheal intubation tube) is successful in approximately 80 to 90% of resuscitation patients, 10 to 20% will develop acute respiratory failure (ARF) in the days following extubation . This incidence is higher in the patients most fragile in the respiratory field (obese patients, chronic obstructive pulmonary disease (COPD), elderly, heart failure, postoperative cardio-thoracic and / or abdominal surgery ...) . The management of post-extubation ARF consists of etiological treatment associated with ventilatory support which usually requires the use of new endotracheal intubation to deliver "invasive" artificial ventilation. This invasive ventilation is responsible for excess morbidity and excess mortality . Therefore, it is fundamental for the physician to prevent by all means the occurrence of ARF post-extubation. One of the most important causes of extubation failure is the imbalance between the burden imposed on the respiratory system and its ability to overcome it, leading to gas exchange abnormalities, namely hypoxia and hypercapnia. Ensuring adequate oxygenation is therefore essential after extubation. In ICU, oxygen therapy is commonly used to improve and provide adequate oxygenation .

Obesity, a major public health problem in the industrialized countries, concerns 10 to 20% of resuscitation admissions in France. It is associated with excess morbidity and longer mechanical ventilation time compared to the general population. Effect on mortality is controversial , some studies suggesting a protective or neutral effect of obesity , named "obesity paradox" . At the ventilatory level, several pathophysiological changes are combined and contribute to an increase in the incidence of respiratory complications . Pulmonary volumes are amputated, the Body Mass Index (BMI) being negatively correlated with the functional residual capacity and vital capacity. The compliance of the respiratory system is reduced by the weight of the chest wall. Decreased compliance and increased airway resistance lead to increased respiratory muscle work. All of these pathophysiological changes in the obese patient explain the over-risk of desaturation and ARF in the post-extubation period. In addition to the intrinsic risk factors associated with obesity, the post-extubation period is marked by numerous risk factors for the development of ARF and extubation failure.

However, the exploration of different modern modalities of adequate post-extubation oxygen therapy in obese resuscitation patients to prevent the occurrence of extubation failure or post-extubation ARF has never been studied.

For over 20 years, Non-Invasive Ventilation (NIV) has been an essential modality in the prevention ("preventive NIV") and management ("curative NIV") of respiratory failure in ICU. The advantages of this ventilation modality are: respect for airway defense mechanisms (speech and cough maintenance), elimination of laryngeal and tracheal trauma induced by an intubation tube, improved comfort, reduction of the risk of bronchopulmonary nosocomial infection .

An alternative to NIV is the simple administration of oxygen. Two devices delivering low oxygen flows are commonly used for oxygen therapy after extubation: the Venturi mask and the nasal cannulas. The nasal cannulas are preferred by patients and less likely to be removed, but they can cause discomfort due to dryness of nasal mucosa when oxygen flows greater than 4 L/min are used. The Venturi mask delivers predetermined oxygen concentrations ranging from 24 to 60%, but the mask is generally less comfortable than the nasal cannula and more likely to be displaced or removed . In clinical practice, the Venturi mask is more frequently used after extubation because critically ill patients breathe preferentially through an open mouth rather than the nose.

More recently, a new oxygen therapy device has been marketed. This device (Optiflow®, Fisher & Paykel, New Zealand) of High Flow Nasal Humidified Oxygen Therapy (HFNO) is able to deliver oxygen humidified by nasal cannulas. This system has several theoretical advantages: high flow rates reduce the dilution of inhaled oxygen and allow precise distribution of FiO2 throughout the inspiratory phase by adapting the peak flow rate to the patient. The high oxygen flow can also have a washing effect on the dead space of the nasopharynx. In addition, a flow-dependent effect helps to generate a continuous positive end-expiratory pressure (PEEP) , related to an air entrainment mechanism, which has been documented in healthy volunteers and COPD patients. Finally, the use of a high level of humidity could prevent alterations of the ciliated epithelium of the respiratory tract, maintain the activity of the muco-ciliary system, and facilitate the elimination of secretions . In a study in non-obese patients, HFNO was shown to improve oxygenation compared to the Venturi mask, while reducing respiratory rate, PaCO2 and discomfort in patients receiving oxygen therapy after extubation. These positive effects of HFNO were associated with less interface displacement and less oxygen desaturations than the Venturi mask. A secondary result was that the need for reintubation at 48 h was lower with HFNO than with the Venturi mask (4% vs 21%).

In summary, in order to decrease the incidence of extubation failure (need for reintubation within 48-72h post-extubation) of the most fragile patients (including obese patients), it is recommended in intensive care unit to prophylactically use various ventilatory support strategies and / or oxygenation, among which:

* NIV which allows to deliver an established level of oxygen delivered via ventilatory assistance using two levels of pressure (inspiratory aid + positive expiratory pressure), but intermittently, with duration of sessions dependent on the tolerance of the patient.
* Oxygen therapy, which can be administered in two ways: HFNO or standard oxygen therapy.

3.2 Knowledge gap and research hypothesis In an observational study of 124 patients, EL Sohl et al. compared NIV to standard oxygen to prevent extubation failure, and showed a 16% absolute risk reduction of ARF using NIV compared to standard oxygen following extubation. In 155 post cardiac surgery obese patients, Corley et al. compared HFNO and standard oxygen to prevent extubation failure, without showing any difference.

However, none of these studies compared simultaneously the most recent devices available: NIV, HFNO and standard oxygen, nor their association. HFNO is now often used, and the PEP issued by HFNO is much lower than that issued by the NIV. The opening of the cells and the probable maintenance of the residual functional capacity is less when using HFNO than NIV. Thus, the two oxygenation methods (NIV and HFNO) appear complementary in case of ARF following extubation in obese patients. The benefit of NIV +/- HFNO compared to oxygen (standard oxygen or HFNO) to improve the quality of post-extubation oxygenation of overall ICU obese patients has never been studied.

In this multicenter, randomized, controlled, interventional study in mechanically ventilated obese critically ill patients, we will test the hypothesis that NIV (associated to HFNO or standard oxygen) is superior to oxygen (HFNO or standard oxygen) to prevent the development of ARF in obese extubated patients in intensive care unit.

3.3 Originality and innovative aspects of the study NIV has proven effective in small observational studies in preventing ARF following extubation of obese patients, in ICU or postoperative setting. The control group was standard oxygen therapy, which was the standard of care a few years ago. Nowadays, HFNO is more and more used, and has proven to be non-inferior to NIV in ARF patients following cardiothoracic surgery and in high risk patients after extubation in the ICU. To date no prospective randomized study has compared NIV (alternated with HFNO or standard oxygen) with oxygen therapy (HFNO or standard oxygen) to prevent extubation failure in obese patients. This study would be the first to compare the association of the most recent advances in term of oxygenation and lung recruitment in critically ill patients: NIV, HFNO and standard oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years)
* Subjects must be covered by public health insurance
* Obese patients defined by a body mass index ≥ 30 kg/m²
* Extubation after a length of mechanical ventilation >= 6 hours
* Written informed consent from the patient or proxy (if present) before inclusion or once possible when patient has been included in a context of emergency.

Exclusion Criteria:

* Refusal of study participation or to pursue the study by the patient
* Hypercapnia with a formal indication for NIV (PaCO2 ≥ 50 mmHg, formal indication for NIV)
* Isolated cardiogenic pulmonary edema (formal indication for NIV). Patients with pulmonary edema associated with another ARF etiology can be included.
* Pregnancy or breastfeeding
* Anatomical factors precluding the use of NIV and/or HFNO
* Absence of coverage by the French statutory healthcare insurance system
* Patients with tracheostomy
* Patients with CPAP for obstructive apnea syndrome
* Patients with decision of no-reintubate (limitation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
The failure of the treatment, defined by a composite criteria | 72 hours
  The failure of the treatment, defined by a composite criteria combining the treatment failure, defined as reintubation for mechanical ventilation, switch to the other study treatment, or premature study-treatment discontinuation

SECONDARY OUTCOMES:
Incidence of acute respiratory failure | up to Day 7
  Occurrence of acute respiratory failure
Oxygenation | Up to Day 7
  Oxygenation will be assessed based on the lowest SpO2 value and on PaO2/FiO2 (if available)
Organ failure | Up to Day 7
  Number of organ failures as assessed by the daily SOFA score each day until Day-7
ICU all-cause mortality | up to day 28
Tracheal intubation rate | up to day 28
Length of stay in ICU and in hospital | up to day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Saint Eloi, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 12 months after the main publication
Access Criteria: Data are provided to qualified investigators free of charge. Required documents to request data include a summary of the research plan, request form, and IRB review. Dataset will be shared after careful examination by the study board of investigators.

REFERENCES:
- [Background] De Jong A, Huguet H, Molinari N, Jaber S. Non-invasive ventilation versus oxygen therapy after extubation in patients with obesity in intensive care units: the multicentre randomised EXTUB-OBESE study protocol. BMJ Open. 2022 Jan 19;12(1):e052712. doi: 10.1136/bmjopen-2021-052712. PMID 35045999
- [Background] De Jong A, Bignon A, Stephan F, Godet T, Constantin JM, Asehnoune K, Sylvestre A, Sautillet J, Blondonnet R, Ferrandiere M, Seguin P, Lasocki S, Rolle A, Fayolle PM, Muller L, Pardo E, Terzi N, Ramin S, Jung B, Abback PS, Guerci P, Sarton B, Roze H, Dupuis C, Cousson J, Faucher M, Lemiale V, Cholley B, Chanques G, Belafia F, Huguet H, Futier E, Azoulay E, Molinari N, Jaber S; EXTUB-OBESE trial group. Effect of non-invasive ventilation after extubation in critically ill patients with obesity in France: a multicentre, unblinded, pragmatic randomised clinical trial. Lancet Respir Med. 2023 Jun;11(6):530-539. doi: 10.1016/S2213-2600(22)00529-X. Epub 2023 Jan 21. PMID 36693403
- [Derived] De Jong A, Huguet H, Bignon A, Stephan F, Godet T, Collet L, Asehnoune K, Sylvestre A, Sautillet J, Blondonnet R, Ferrandiere M, Launey Y, Lasocki S, Rolle A, Fayolle PM, Muller L, Pardo E, Terzi N, Ramin S, Jung B, Weiss E, Abback PS, Guerci P, Sarton B, Roze H, Dupuis C, Cousson J, Faucher M, Lemiale V, Cholley B, Chanques G, Belafia F, Chauveton C, Futier E, Azoulay E, Molinari N, Jaber S; EXTUB-OBESE trial group. Noninvasive ventilation in postoperative critically ill patients with morbid obesity: secondary analysis of the EXTUBOBESE multicentre randomised clinical trial. Br J Anaesth. 2025 Nov;135(5):1477-1485. doi: 10.1016/j.bja.2025.09.002. Epub 2025 Oct 3. PMID 41046173
- [Derived] De Jong A, Capdevila M, Aarab Y, Rabboni F, Kozoriz A, Heupel G, Pensier J, Lakbar I, Monet C, Chanques G, Jaber S. Norepinephrine use at extubation in critically ill patients with obesity: a cohort study with multicenter validation. Intensive Care Med. 2025 Dec;51(12):2341-2353. doi: 10.1007/s00134-025-08066-x. Epub 2025 Aug 6. PMID 40768069